CLINICAL TRIAL: NCT00660478
Title: Randomized Clinical Comparison of the Endeavor and the Cypher Coronary Stents in Non-selected Angina Pectoris Patients
Acronym: SORT-OUTIII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Evald Hoej Christiansen (Other)
Collaborators: Aalborg University Hospital (Other); Odense University Hospital (Other); University Hospital, Gentofte, Copenhagen (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Evald Hoej Christiansen, MD, Aarhus University Hospital Skejby
Organization: Aarhus University Hospital Skejby (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 20050194
Record Dates: First submitted 2008-04-09; First posted 2008-04-17 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2008-09

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Zotarolimus eluting stent
  Interventions: Device: Endeavor
- 2 (Active Comparator): Sirolimus stent
  Interventions: Device: Cypher Select

INTERVENTIONS:
Device: Endeavor — Comparison of two different drug eluting coronary stents
  Other Names: 1. Endeavor
  Arms: 1
Device: Cypher Select — Comparison of two different drug eluting coronary stents
  Other Names: 1. Cypher
  Arms: 2

SUMMARY:
Randomized clinical comparison of the serolimus eluting Cypher stent and the zotarolimus eluting Endeavor stent.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated with one or more drug eluting stents in the coronary arteries at one of the 5 heart centers in Denmark can be included in the study.

Exclusion Criteria:

* The patient will not participate
* The patient participates in other randomized stent studies
* Expected survival < 1 year
* Allergy to Aspirin, Clopidogrel or Ticlopidine
* Allergy to Sirolimus or ABT-578

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2342 (Actual)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
In a randomized study to compare the Endeavor and the Cypher Select coronary stents by assessing MACE (cardiac death, myocardial infarction, stent thrombosis and target vessel revascularization) after 9 months. | 9 months

SECONDARY OUTCOMES:
To compare device success rate, procedure success rate and complication rate during hospitalization, after 1 month and after 9 months. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Jens F Lassen, MD, PhD, Study Chair — Aarhus University Hospital Skejby; Klaus Rasmussen, MD, DMSc, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aarhus University Hospital, Skejby, Aarhus, Denmark

REFERENCES:
- [Derived] Maeng M, Tilsted HH, Jensen LO, Krusell LR, Kaltoft A, Kelbaek H, Villadsen AB, Ravkilde J, Hansen KN, Christiansen EH, Aaroe J, Jensen JS, Kristensen SD, Botker HE, Thuesen L, Madsen M, Thayssen P, Sorensen HT, Lassen JF. Differential clinical outcomes after 1 year versus 5 years in a randomised comparison of zotarolimus-eluting and sirolimus-eluting coronary stents (the SORT OUT III study): a multicentre, open-label, randomised superiority trial. Lancet. 2014 Jun 14;383(9934):2047-2056. doi: 10.1016/S0140-6736(14)60405-0. Epub 2014 Mar 14. PMID 24631162
- [Derived] Maeng M, Tilsted HH, Jensen LO, Kaltoft A, Kelbaek H, Abildgaard U, Villadsen AB, Krusell LR, Ravkilde J, Hansen KN, Christiansen EH, Aaroe J, Jensen JS, Kristensen SD, Botker HE, Madsen M, Thayssen P, Sorensen HT, Thuesen L, Lassen JF. 3-Year clinical outcomes in the randomized SORT OUT III superiority trial comparing zotarolimus- and sirolimus-eluting coronary stents. JACC Cardiovasc Interv. 2012 Aug;5(8):812-8. doi: 10.1016/j.jcin.2012.04.008. PMID 22917452
- [Derived] Jensen LO, Maeng M, Thayssen P, Villadsen A, Krusell L, Botker HE, Pedersen KE, Aaroe J, Christiansen EH, Vesterlund T, Hansen KN, Ravkilde J, Tilsted HH, Lassen JF, Thuesen L. Late lumen loss and intima hyperplasia after sirolimus-eluting and zotarolimus-eluting stent implantation in diabetic patients: the diabetes and drug-eluting stent (DiabeDES III) angiography and intravascular ultrasound trial. EuroIntervention. 2011 Jul;7(3):323-31. doi: 10.4244/EIJV7I3A56. PMID 21729834
- [Derived] Rasmussen K, Maeng M, Kaltoft A, Thayssen P, Kelbaek H, Tilsted HH, Abildgaard U, Christiansen EH, Engstrom T, Krusell LR, Ravkilde J, Hansen PR, Hansen KN, Abildstrom SZ, Aaroe J, Jensen JS, Kristensen SD, Botker HE, Madsen M, Johnsen SP, Jensen LO, Sorensen HT, Thuesen L, Lassen JF; SORT OUT III study group. Efficacy and safety of zotarolimus-eluting and sirolimus-eluting coronary stents in routine clinical care (SORT OUT III): a randomised controlled superiority trial. Lancet. 2010 Mar 27;375(9720):1090-9. doi: 10.1016/S0140-6736(10)60208-5. Epub 2010 Mar 16. PMID 20231034